CLINICAL TRIAL: NCT05832632
Title: A Randomized Controlled Trial Comparing 3 Formats of Mindfulness Interventions to an Active Control Intervention in a Population With Elevated Levels of Stress: Effects of Subjective and Physiological Stress
Brief Title: The Effect of Mindfulness on Psychophysiological Stress in a Population With Elevated Stress Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Headspace Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 45345
Record Dates: First submitted 2023-03-30; First posted 2023-04-27 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Psychological Stress; Physiological Stress
Keywords: Stress; Mindfulness; HRV
MeSH Terms: conditions — Stress, Psychological | interventions — Sound Recordings

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Headspace Basics Program (Experimental)
  Interventions: Behavioral: Headspace Basics Program
- Headspace Breathing Exercises (Experimental)
  Interventions: Behavioral: Headspace Breathing Exercises
- Headspace Stress Program (Experimental)
  Interventions: Behavioral: Headspace Stress Program
- Active Control (Audiobook) (Active Comparator)
  Interventions: Behavioral: Active Control (Audiobook)
- Passive Control (No Intervention)

INTERVENTIONS:
Behavioral: Headspace Basics Program — 30-day smartphone-based mindfulness intervention consisting of 10 minutes per day. The program consist of generic mindfulness techniques such as breath awareness, body scans, mindful noting of thoughts and emotions.
  Arms: Headspace Basics Program
Behavioral: Headspace Breathing Exercises — 30-day smartphone-based breathing exercises. Each exercise consists of box breathing for 1 minute and participants are instructed to complete 10 sessions corresponding to 10 minutes per day.
  Arms: Headspace Breathing Exercises
Behavioral: Headspace Stress Program — 20-day smartphone-based mindfulness intervention consisting of 15 minutes per day. The Stress program content is based on well-established concepts and practices within stress management, and mindfulness, and is targeted to people with elevated stress.
  Arms: Headspace Stress Program
Behavioral: Active Control (Audiobook) — 30-day smartphone-based Audiobook book consisting of 10 minutes per day.
  Arms: Active Control (Audiobook)

SUMMARY:
Stress-related disorders have over the last decade increased and contributed to a worldwide disease burden. At the same time there is limited treatment access for mental health disorders, which has left many people without necessary care. However, in recent years there has been a rise in digital mindfulness interventions. Specifically, these interventions have focused on smartphone-based applications as an effective format for mindfulness training programs. Thus, the goal of this randomized controlled trial is to test the effects of three types of mindfulness programs in a population with elevated stress. The three formats of mindfulness interventions are identical in total training duration but varies in content and intervention length. Specifically, the first intervention consists of programmatic mindfulness content that progress over the course of 30 sessions with a duration of 10 min per session. The second intervention consists of single succinct breathing exercises with no programmatic content over the course of 30 sessions with a duration of 10 min per session. The third intervention consists of mindfulness-based content specifically targeted to people with elevated stress that progress over the course of 20 sessions with a duration of 15 min per session. An active control group listening to an audiobook over the course of 30 sessions with a duration of 10 min per session will be employed and a passive control group.

The study will evaluate outcomes related to subjective stress, sleep quality, mindfulness and physiological effects of stress using HRV.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to high perceived stress based on PSS total scores (14-40)
* Fluent in English

Exclusion Criteria:

* Regular mindfulness practice for more than 1 month within the last year
* Medical diagnosis e.g. psychiatric/neurological conditions
* Low levels of stress (i.e., less than a score of 14 assessed with the PSS)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 225 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS-10) | immediately post intervention
Heart rate variability (HRV) | immediately post intervention
  HRV data will be recorded continuously during a rest period, acute stress period*, and recovery period at both pre and post on a subject-by-subject basis.
  *The study will use an acute stress manipulation, specifically the CPT (Cold Pressor Task). The CPT is a standardized physiological acute stressor which has been shown to induce stress, reflected in autonomic stress reactivity (e.g. Lupien et al., 2007; Raio et al., 2017).

SECONDARY OUTCOMES:
The Pittsburgh Sleep Quality Index (PSQI) | immediately post intervention
Mindful Attention Awareness Scale (MAAS) | immediately post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Kirk, PhD, Principal Investigator — University of Southern Denmark
Locations (1):
- University of Southern Denmark. Department of Psychology., Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen, S., & Janicki-Deverts, D. (2012), Who's Stressed? Distributions of Psychological Stress in the United States in Probability Samples from 1983, 2006, and 2009. Journal of Applied Social Psychology, 42: 1320-1334. https://doi.org/10.1111/j.1559-1816.2012.00900.x
- [Background] Tian F, Shen Q, Hu Y, Ye W, Valdimarsdottir UA, Song H, Fang F. Association of stress-related disorders with subsequent risk of all-cause and cause-specific mortality: A population-based and sibling-controlled cohort study. Lancet Reg Health Eur. 2022 May 28;18:100402. doi: 10.1016/j.lanepe.2022.100402. eCollection 2022 Jul. PMID 35663363
- [Background] World Health Organization. The impact of COVID-19 on mental, neurological and substance use services: results of rapid assessment. Geneva: World Health Organization; 2020. Available from: https://www.who.int/publications-detail-redirect/978924012455
- [Background] Sorkin DH, Janio EA, Eikey EV, Schneider M, Davis K, Schueller SM, Stadnick NA, Zheng K, Neary M, Safani D, Mukamel DB. Rise in Use of Digital Mental Health Tools and Technologies in the United States During the COVID-19 Pandemic: Survey Study. J Med Internet Res. 2021 Apr 16;23(4):e26994. doi: 10.2196/26994. PMID 33822737
- [Background] Philippe TJ, Sikder N, Jackson A, Koblanski ME, Liow E, Pilarinos A, Vasarhelyi K. Digital Health Interventions for Delivery of Mental Health Care: Systematic and Comprehensive Meta-Review. JMIR Ment Health. 2022 May 12;9(5):e35159. doi: 10.2196/35159. PMID 35551058
- [Background] Raio CM, Hartley CA, Orederu TA, Li J, Phelps EA. Stress attenuates the flexible updating of aversive value. Proc Natl Acad Sci U S A. 2017 Oct 17;114(42):11241-11246. doi: 10.1073/pnas.1702565114. Epub 2017 Oct 2. PMID 28973957
- [Background] Lupien SJ, Maheu F, Tu M, Fiocco A, Schramek TE. The effects of stress and stress hormones on human cognition: Implications for the field of brain and cognition. Brain Cogn. 2007 Dec;65(3):209-37. doi: 10.1016/j.bandc.2007.02.007. Epub 2007 Apr 26. PMID 17466428
- [Derived] Kirk U, Staiano W, Hu E, Ngnoumen C, Kunkle S, Shih E, Clausel A, Purvis C, Lee L. App-Based Mindfulness for Attenuation of Subjective and Physiological Stress Reactivity in a Population With Elevated Stress: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2023 Oct 13;11:e47371. doi: 10.2196/47371. PMID 37831493